CLINICAL TRIAL: NCT06793722
Title: The Effect of Technological Devices on the Child's Pain and Anxiety Level in Circumcision Performed With Local Anesthesia
Brief Title: Technological Devices in Circumcision
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University (Other)
Responsible Party: Principal Investigator, Bedreddin Kalyenci, Principal Investigator, Adiyaman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HRÜ/24.21.25
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Circumcision Adult; Circumcision, Male; Circumcision
Keywords: circumcision
MeSH Terms: interventions — Circumcision, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- circumcision by watching videos/playing games (Experimental)
  Interventions: Procedure: Technological device in circumcision
- circumcision without visual or verbal stimulation (No Intervention): Not providing any visual or verbal stimulation to circumcised children

INTERVENTIONS:
Procedure: Technological device in circumcision — Circumcision is performed by watching a video/playing a game during the procedure in children who are circumcised.
  Arms: circumcision by watching videos/playing games

SUMMARY:
It aims to investigate the effect of circumcision on the pain and anxiety level of children who are circumcised by watching videos/playing games during the procedure. Previous studies have been conducted to explain the procedure with informative videos and games before circumcision, and reductions in anxiety and pain levels have been detected. The research will start with hospitalization and end with a check-up after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Circumcision for medical or religious reasons.

Exclusion Criteria:

* Children with chronic diseases.
* Children with genital medical problems.
* Children with mental and communication disabilities and their parents.

Ages: 6 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
change of child anxiety and worry | immediately after the intervention/procedure/surgery
  Anxiety levels will be assessed with scales to determine changes in anxiety.
  Wong Baker Facial Pain Scale:
  " 0 " Very happy because no pain, " 1 " A little pain, " 2 " A little more pain, " 3 " More pain, " 4 " Quite a lot of pain, " 5 " The worst pain you can imagine. Situational Anxiety Scale: The scale, which has been translated into Turkish and adapted, consists of a total of 20 items. The highest score that can be obtained from the scale is 80, and the lowest is 20.
  Child fear scale:This scale includes 5 different facial expressions. This scale is scored between 0-4.

SECONDARY OUTCOMES:
Changes in anxiety and worry among parents. | immediately after the intervention/procedure/surgery
  Anxiety levels will be assessed with scales to determine changes in anxiety. The Beck Anxiety Inventory (BAI) consists of 21 self-reported items (four-point scale) used to assess the intensity of physical and cognitive anxiety symptoms during the past week. Scores may range from 0 to 63: minimal anxiety levels (0-7), mild anxiety (8-15), moderate anxiety (16-25), and severe anxiety (26-63).

CONTACTS AND LOCATIONS:
Locations (1):
- Adıyaman University, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 2 years after completion of the work